CLINICAL TRIAL: NCT02838485
Title: Cortical Activation in Individuals With Finger Amputation During Mirror Versus Imagery Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Mirror- HMO-CTIL
Record Dates: First submitted 2016-07-17; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Amputees

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amputees (Experimental): The subjects will receive both mirror and imagery treatments in a cross-over design.
  Interventions: Other: Mirror; Other: Imagery

INTERVENTIONS:
Other: Mirror — The healthy hand will be mirrored and the amputated hand unseen by the subject while performing hand movements.
Other: Imagery — The subject will be asked to imagine performing hand movements.

SUMMARY:
Goals : ( a) to examine differences in cortical activity during hand movements with a mirror compared to imagery of the same movements, and (b) to examine correlation between cortical activity during imagery or mirror treatment and the pain and performance measures in finger amputees.

A cross-sectional study of 20 subjects in a Functional Magnetic Resonance Imaging (fMRI) preforming mirror therapy hand movement and imagery hand movement. Also, Visual Analogue Scale for pain and the Disability of the Arm, Shoulder and Hand (DASH) questionnaire and Jebsen Taylor Hand Function Test will be used.

DETAILED DESCRIPTION:
Goals : ( a) to examine differences in cortical activity during hand movements with a mirror compared to imagery of the same movements, and (b) to examine correlation between cortical activity during imagery or mirror treatment and the pain and performance measures in finger amputees.

A cross-sectional one-meeting study of 20 subjects (finger amputees) in a Functional Magnetic Resonance Imaging (fMRI) preforming mirror therapy hand movement and imagery hand movement. Also, Visual Analogue Scale for pain and the Disability of the Arm, Shoulder and Hand (DASH) questionnaire and Jebsen Taylor Hand Function Test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Following unilateral traumatic finger or fingers amputation (1 to 3 fingers)
* Self-reported limited functionality, sensory disorder or pain

Exclusion Criteria:

* Are not comparable with MRI restrictions
* Chronic pain disease
* Psychiatric condition

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Cortical activity | 1 hour
  Activation of supplementary motor area (SMA), S1 and M1.

SECONDARY OUTCOMES:
Visual analogue scale | 10 minutes
  Filled by the subject for subjective pain in residuum discomfort.
Disability of the Arm, Shoulder and Hand | 30 minutes
  Questionnaire regarding the disability and daily activities difficulties.
The Jebsen Taylor Hand Function Test | 30 minutes
  Standard evaluation of hands functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Chan BL, Witt R, Charrow AP, Magee A, Howard R, Pasquina PF, Heilman KM, Tsao JW. Mirror therapy for phantom limb pain. N Engl J Med. 2007 Nov 22;357(21):2206-7. doi: 10.1056/NEJMc071927. No abstract available. PMID 18032777
- [Background] Deconinck FJ, Smorenburg AR, Benham A, Ledebt A, Feltham MG, Savelsbergh GJ. Reflections on mirror therapy: a systematic review of the effect of mirror visual feedback on the brain. Neurorehabil Neural Repair. 2015 May;29(4):349-61. doi: 10.1177/1545968314546134. Epub 2014 Aug 26. PMID 25160567